CLINICAL TRIAL: NCT02366429
Title: Psychological Treatment Via the Internet for Antenatal Depression
Brief Title: ICBT for Antenatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Viktor Kaldo, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20141959311
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Antenatal Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICBT (Experimental): Internet-based CBT for antenatal depression
  Interventions: Behavioral: ICBT for antenatal depression
- TAU (Active Comparator): Treatment as usual provided at antenatal clinics and other health care instances
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: ICBT for antenatal depression — Participants receives active therapist support via the internet to go through a 10-week self-help treatment on a secure web platform
  Arms: ICBT
Other: TAU — Treatment as usual provided at antenatal clinics and other health care instances
  Arms: TAU

SUMMARY:
Randomized controlled trial evaluating an Internet-delivered Cognitive Behavioral Therapy (ICBT) adapted for pregnant women suffering from antenatal depression. The ICBT-program will be added to treatment as usual (TAU) and compared to TAU only.

Participants (n=60) are recruited from all over Sweden (only Swedish citizens can participate) and are assessed and treated on a distance via a secure web platform and telephone.

DETAILED DESCRIPTION:
In order to evaluate feasibility and effectiveness of an ICBT-program for antenatal depression that will be used in a larger clinical trial, the current RCT (n=60) will be performed and act as a pilot for the main study.

Participants will all be receiving the regular treatment (TAU) provided at their antenatal clinic and other health care instances. Half of them will be randomized to an add-on of a previously established 10-week long ICBT-program for depression in general, now adapted for pregnant women. The other half will receive TAU during 10 weeks and then freely decide if they want to participate in the pregnancy-adapted ICBT-program (only possible if 10 or more weeks left till estimated delivery date), start the regular ICBT-program for depression within 2-6 weeks post-partum, or decline ICBT-treatment. The participants in this study will be recruited from all over Sweden via internet, advertisements and information at antenatal clinics. A web-based screening questionnaire will form the basis for a first assessment and review of inclusion criteria, followed by a structured telephone interview where diagnoses (SCID-1 for depression, adjusted for DSM 5, and M.I.N.I. for other diagnoses and assessment of suicide risk) and suitability will be assessed, a CGI-rating will be performed, and the final decision on inclusion will be made.

Level of depression pre- and post-treatment will be assessed with MADRS-S filled out via the internet-treatment platform together with the other self-rating measures used in the main study. A questionnaire where the participants evaluate the content of the adapted ICBT-program and their own use and perceived benefit of the treatment methods will also be given at post-treatment and during treatment.

Structured telephone interview will be held at post-treatment, primarily to assess the content of TAU, to administer CGI and a standardized version for MADRS-S (designed to replace missing questionnaire data), and to make a qualitative evaluation of the participants view of the adapted ICBT-program.

The estimated effect of ICBT compared to TAU is 0.8 (Cohen's d) and with 60 participants and some attrition this will result in a statistical power of 80% for this initial, smaller RCT.

ELIGIBILITY:
Inclusion Criteria:

* pregnant female > 18 years old at gestational week 11-28
* verified moderate depression according to SCID-I with or without concomitant anxiety disorder
* able to understand the Swedish language orally and in written
* able to use the internet for the ICBT
* currently in contact with an antenatal clinic to receive regular care

Exclusion Criteria:

* known drug or alcohol abuse
* serious somatic disorder or psychiatric disorder such as psychosis, bipolar disorder, severe personality disorder, autism or mental retardation and severe melancholic or psychotic depression,
* having started or changed medication with SSRI, SNRI or mood-stabilizers within 3 weeks,
* according to psychiatric assessment have a high suicide risk will be excluded from the study. These women will be helped to receive necessary psychiatric treatment as usual.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Self-rated depression measured by Montgomery Asberg Depression Rating Scale | Change from baseline to post-treatment (after 10 weeks) and to 3-4 weeks post-partum
  Depression measured by Montgomery Asberg Depression Rating Scale (MADRS-S), a 9-item self-rated measure of change in depression severity. It also screens for suicidality.

SECONDARY OUTCOMES:
Self-rated antenatal depression Edinburgh Postnatal Depression Scale | Change from baseline to post-treatment (after 10 weeks) and to 3-4 weeks post-partum
  Edinburgh Postnatal Depression Scale (EPDS; Cox, Holden & Sagovsky, 1987)
Self-rated function Work and Social Adjustment Scale | Change from baseline to post-treatment (after 10 weeks) and to 3-4 weeks post-partum
  Work and Social Adjustment Scale (WSAS; Zahra et al., 2014)
Self-rated Insomnia Insomnia Severity Index | Change from baseline to post-treatment (after 10 weeks) and to 3-4 weeks post-partum
  Insomnia Severity Index (ISI; Bastien, Vallieres & Morin, 2001)
Self-rated function/quality of life Euroqol | Change from baseline to post-treatment (after 10 weeks) and to 3-4 weeks post-partum
  Euroqol (EQ-5D ; Hinz et al., 2006),
Self-rated anxiety and worry GAD-7 | Change from baseline to post-treatment (after 10 weeks) and to 3-4 weeks post-partum
  GAD-7(Beard, & Björgvinsson, 2014)
Expert rating of overall disease burden Clinical Global Impression - Severity scale | Change from baseline to post-treatment (after 10 weeks) and to 3-4 weeks post-partum
  Clinical Global Impression - Severity scale (CGI-S; Guy, 2000)

CONTACTS AND LOCATIONS:
Locations (1):
- Internetpsykiatrienehten (Internet Psychiatry Unit), Psykiatri Sydväst, SLSO, Stockholm, Sweden

REFERENCES:
- [Derived] Forsell E, Bendix M, Hollandare F, Szymanska von Schultz B, Nasiell J, Blomdahl-Wetterholm M, Eriksson C, Kvarned S, Lindau van der Linden J, Soderberg E, Jokinen J, Wide K, Kaldo V. Internet delivered cognitive behavior therapy for antenatal depression: A randomised controlled trial. J Affect Disord. 2017 Oct 15;221:56-64. doi: 10.1016/j.jad.2017.06.013. Epub 2017 Jun 13. PMID 28628768
- See also: Related Info — http://www.internetpsykiatri.se